CLINICAL TRIAL: NCT05693376
Title: Evaluation of a Screening Algorithm for Early Detection of Occult Cardiac Amyloidosis in Subjects at Risk
Brief Title: Screening Algorithm for Early Detection of Occult Cardiac Amyloidosis
Acronym: EARLY-CA
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Maria Papathanasiou, Principal Investigator, Cardiologist, University Hospital, Essen
Other Study IDs: 209268
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Amyloidosis
Keywords: Cardiac amyloidosis; Aortic stenosis; AS-ATTR
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Subjects who meet the following inclusion criteria: 1) Severe aortic stenosis. 2) Age > 65 years for male and >70 years for female. 3) Increased left ventricular wall thickness ≥14 mm. 4) Blood pressure ≤ 140/90 mmHg and at least 1 major or ≥ 2 minor criteria. Major criteria: a) Carpal tunnel syndrom; b) Non-traumatic rupture of the biceps tendon; c) NT-proBNP > 1000 pg/ml; d) hs Troponin value above the 99th percentile without dynamic changes (≤ 20%). Minor criteria: a) Diastolic dysfunction (at least grade 2, E' < 10 cm/s); b) Sinus bradycardia/AV block/pacemaker; c) Atrial fibrillation.
- Control group: Subjects who meet the following inclusion criteria: 1) Severe aortic stenosis. 2) Age > 65 years for male and >70 years for female. 3) Increased left ventricular wall thickness ≥14 mm. 4) Blood pressure ≤ 140/90 mmHg.

SUMMARY:
Early diagnosis of cardiac amyloidosis (CA) is crucial because of the poor overall survival, high mortality and the need for early therapy including new treatment possibilities for transthyretin amyloidosis. Previously considered a rare condition, CA is being demonstrated to account for up to 17 % of heart failure with preserved ejection fraction cases as well as up to 16 % of Patients with severe aortic stenosis, undergoing surgical of transcatheter aortic valve replacement. It seems that CA is being underdiagnosed as the data of post-mortem studies demonstrate that at least 25% of elderly individuals have histologic evidence of amyloid deposits. Other common conditions with increased afterload such as hypertensive or hypertrophic heart disease that mimic echocardiographic features or clinical symptoms may be the reason of postponed recognition of CA. Furthermore, the lack of definitive biomarkers makes the diagnosis even more challenging. However, it has been shown that some clinical, laboratory and echocardiographic findings, so called "red flags", may indicate occult CA. A deeper and constructive analysis of the findings and establishment of prediction criteria could possibly lead to improvement of early CA recognition and survival in subjects at risk. We aim to prospectively perform a systematic screening for CA in individuals at risk based on predefined selection criteria. Our aim is to evaluate if specific criteria would lead to increased detection of CA and in this case, to define major and minor diagnostic criteria.

DETAILED DESCRIPTION:
The study aims to perform a prospective screening and detect occult CA in subjects at risk with aortic valve stenosis, undergoing either transcatheter or surgical aortic valve replacement. The study has two main objectives. Firstly, we aim to determine the real prevalence of CA according to the targeted "red flags" analysis and secondly, we aim to establish an algorithm for early detection of CA.

ELIGIBILITY:
Inclusion Criteria:

* Fulfillment of following four criteria: 1) Severe aortic stenosis. 2) Age > 65 years for male and >70 years for female. 3) Increased left ventricular wall thickness ≥14 mm. 4) Blood pressure ≤ 140/90 mmHg and at least 1 major or ≥ 2 minor criteria.

Major criteria:

1. Carpal tunnel syndrom
2. Non-traumatic rupture of the biceps tendon
3. NT-proBNP > 1000 pg/ml
4. hs Troponin value above the 99th percentile without dynamic changes (≤ 20%)

Minor criteria:

1. Diastolic dysfunction (at least grade 2, E' < 10 cm/s)
2. Sinus bradycardia/AV block/pacemaker
3. Atrial fibrillation

Exclusion Criteria:

* Known cardiac amyloidosis (ATTR or AL)
* Unable to provide written informed consent
* Refusal to provide written informed consent
* Contraindications for study investigations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with severe aortic stenosis, that fulfill the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Diagnosis of occult cardiac amyloidosis | 3 years
  Early diagnosis of occult cardiac amyloidosis, based on a proposed screening algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Aiste Monika Jakstaite, MD, Principal Investigator — University Hospital, Essen
Locations (1):
- University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maurer MS, Elliott P, Comenzo R, Semigran M, Rapezzi C. Addressing Common Questions Encountered in the Diagnosis and Management of Cardiac Amyloidosis. Circulation. 2017 Apr 4;135(14):1357-1377. doi: 10.1161/CIRCULATIONAHA.116.024438. PMID 28373528
- [Background] Gonzalez-Lopez E, Gallego-Delgado M, Guzzo-Merello G, de Haro-Del Moral FJ, Cobo-Marcos M, Robles C, Bornstein B, Salas C, Lara-Pezzi E, Alonso-Pulpon L, Garcia-Pavia P. Wild-type transthyretin amyloidosis as a cause of heart failure with preserved ejection fraction. Eur Heart J. 2015 Oct 7;36(38):2585-94. doi: 10.1093/eurheartj/ehv338. Epub 2015 Jul 28. PMID 26224076
- [Background] Fajardo J, Cummings A, Brown E, Cuomo K, Rhodes P, Woodbury S, Gilotra N, Russell S, Judge D. Clinical pathway to screen for cardiac amyloidosis in heart failure with preserved ejection fraction. Amyloid. 2019;26(sup1):166-167. doi: 10.1080/13506129.2019.1583178. No abstract available. PMID 31343333
- [Background] Mohammed SF, Mirzoyev SA, Edwards WD, Dogan A, Grogan DR, Dunlay SM, Roger VL, Gertz MA, Dispenzieri A, Zeldenrust SR, Redfield MM. Left ventricular amyloid deposition in patients with heart failure and preserved ejection fraction. JACC Heart Fail. 2014 Apr;2(2):113-22. doi: 10.1016/j.jchf.2013.11.004. PMID 24720917
- [Background] Longhi S, Lorenzini M, Gagliardi C, Milandri A, Marzocchi A, Marrozzini C, Saia F, Ortolani P, Biagini E, Guidalotti PL, Leone O, Rapezzi C. Coexistence of Degenerative Aortic Stenosis and Wild-Type Transthyretin-Related Cardiac Amyloidosis. JACC Cardiovasc Imaging. 2016 Mar;9(3):325-7. doi: 10.1016/j.jcmg.2015.04.012. Epub 2015 Jul 15. No abstract available. PMID 26189123
- [Background] Treibel TA, Fontana M, Gilbertson JA, Castelletti S, White SK, Scully PR, Roberts N, Hutt DF, Rowczenio DM, Whelan CJ, Ashworth MA, Gillmore JD, Hawkins PN, Moon JC. Occult Transthyretin Cardiac Amyloid in Severe Calcific Aortic Stenosis: Prevalence and Prognosis in Patients Undergoing Surgical Aortic Valve Replacement. Circ Cardiovasc Imaging. 2016 Aug;9(8):e005066. doi: 10.1161/CIRCIMAGING.116.005066. PMID 27511979
- [Background] Castano A, Narotsky DL, Hamid N, Khalique OK, Morgenstern R, DeLuca A, Rubin J, Chiuzan C, Nazif T, Vahl T, George I, Kodali S, Leon MB, Hahn R, Bokhari S, Maurer MS. Unveiling transthyretin cardiac amyloidosis and its predictors among elderly patients with severe aortic stenosis undergoing transcatheter aortic valve replacement. Eur Heart J. 2017 Oct 7;38(38):2879-2887. doi: 10.1093/eurheartj/ehx350. PMID 29019612
- [Background] Cornwell GG 3rd, Murdoch WL, Kyle RA, Westermark P, Pitkanen P. Frequency and distribution of senile cardiovascular amyloid. A clinicopathologic correlation. Am J Med. 1983 Oct;75(4):618-23. doi: 10.1016/0002-9343(83)90443-6. PMID 6624768
- [Background] Tanskanen M, Peuralinna T, Polvikoski T, Notkola IL, Sulkava R, Hardy J, Singleton A, Kiuru-Enari S, Paetau A, Tienari PJ, Myllykangas L. Senile systemic amyloidosis affects 25% of the very aged and associates with genetic variation in alpha2-macroglobulin and tau: a population-based autopsy study. Ann Med. 2008;40(3):232-9. doi: 10.1080/07853890701842988. PMID 18382889
- [Background] Lee MH, Lee SP, Kim YJ, Sohn DW. Incidence, diagnosis and prognosis of cardiac amyloidosis. Korean Circ J. 2013 Nov;43(11):752-60. doi: 10.4070/kcj.2013.43.11.752. Epub 2013 Nov 30. PMID 24363751
- [Background] Desport E, Bridoux F, Sirac C, Delbes S, Bender S, Fernandez B, Quellard N, Lacombe C, Goujon JM, Lavergne D, Abraham J, Touchard G, Fermand JP, Jaccard A; Centre national de reference pour l'amylose AL et les autres maladies par depots d'immunoglobulines monoclonales. Al amyloidosis. Orphanet J Rare Dis. 2012 Aug 21;7:54. doi: 10.1186/1750-1172-7-54. PMID 22909024
- [Background] Maurer MS, Schwartz JH, Gundapaneni B, Elliott PM, Merlini G, Waddington-Cruz M, Kristen AV, Grogan M, Witteles R, Damy T, Drachman BM, Shah SJ, Hanna M, Judge DP, Barsdorf AI, Huber P, Patterson TA, Riley S, Schumacher J, Stewart M, Sultan MB, Rapezzi C; ATTR-ACT Study Investigators. Tafamidis Treatment for Patients with Transthyretin Amyloid Cardiomyopathy. N Engl J Med. 2018 Sep 13;379(11):1007-1016. doi: 10.1056/NEJMoa1805689. Epub 2018 Aug 27. PMID 30145929
- [Background] Solomon SD, Adams D, Kristen A, Grogan M, Gonzalez-Duarte A, Maurer MS, Merlini G, Damy T, Slama MS, Brannagan TH 3rd, Dispenzieri A, Berk JL, Shah AM, Garg P, Vaishnaw A, Karsten V, Chen J, Gollob J, Vest J, Suhr O. Effects of Patisiran, an RNA Interference Therapeutic, on Cardiac Parameters in Patients With Hereditary Transthyretin-Mediated Amyloidosis. Circulation. 2019 Jan 22;139(4):431-443. doi: 10.1161/CIRCULATIONAHA.118.035831. PMID 30586695
- [Background] Witteles RM, Bokhari S, Damy T, Elliott PM, Falk RH, Fine NM, Gospodinova M, Obici L, Rapezzi C, Garcia-Pavia P. Screening for Transthyretin Amyloid Cardiomyopathy in Everyday Practice. JACC Heart Fail. 2019 Aug;7(8):709-716. doi: 10.1016/j.jchf.2019.04.010. Epub 2019 Jul 10. PMID 31302046
- [Background] Oerlemans MIFJ, Rutten KHG, Minnema MC, Raymakers RAP, Asselbergs FW, de Jonge N. Cardiac amyloidosis: the need for early diagnosis. Neth Heart J. 2019 Nov;27(11):525-536. doi: 10.1007/s12471-019-1299-1. PMID 31359320
- [Background] Geller HI, Singh A, Alexander KM, Mirto TM, Falk RH. Association Between Ruptured Distal Biceps Tendon and Wild-Type Transthyretin Cardiac Amyloidosis. JAMA. 2017 Sep 12;318(10):962-963. doi: 10.1001/jama.2017.9236. PMID 28898370
- [Background] Damy T, Costes B, Hagege AA, Donal E, Eicher JC, Slama M, Guellich A, Rappeneau S, Gueffet JP, Logeart D, Plante-Bordeneuve V, Bouvaist H, Huttin O, Mulak G, Dubois-Rande JL, Goossens M, Canoui-Poitrine F, Buxbaum JN. Prevalence and clinical phenotype of hereditary transthyretin amyloid cardiomyopathy in patients with increased left ventricular wall thickness. Eur Heart J. 2016 Jun 14;37(23):1826-34. doi: 10.1093/eurheartj/ehv583. Epub 2015 Nov 3. PMID 26537620
- [Background] Grogan M, Scott CG, Kyle RA, Zeldenrust SR, Gertz MA, Lin G, Klarich KW, Miller WL, Maleszewski JJ, Dispenzieri A. Natural History of Wild-Type Transthyretin Cardiac Amyloidosis and Risk Stratification Using a Novel Staging System. J Am Coll Cardiol. 2016 Sep 6;68(10):1014-20. doi: 10.1016/j.jacc.2016.06.033. PMID 27585505
- [Background] Rapezzi C, Quarta CC, Guidalotti PL, Longhi S, Pettinato C, Leone O, Ferlini A, Salvi F, Gallo P, Gagliardi C, Branzi A. Usefulness and limitations of 99mTc-3,3-diphosphono-1,2-propanodicarboxylic acid scintigraphy in the aetiological diagnosis of amyloidotic cardiomyopathy. Eur J Nucl Med Mol Imaging. 2011 Mar;38(3):470-8. doi: 10.1007/s00259-010-1642-7. Epub 2010 Nov 11. PMID 21069320
- [Background] Gillmore JD, Maurer MS, Falk RH, Merlini G, Damy T, Dispenzieri A, Wechalekar AD, Berk JL, Quarta CC, Grogan M, Lachmann HJ, Bokhari S, Castano A, Dorbala S, Johnson GB, Glaudemans AW, Rezk T, Fontana M, Palladini G, Milani P, Guidalotti PL, Flatman K, Lane T, Vonberg FW, Whelan CJ, Moon JC, Ruberg FL, Miller EJ, Hutt DF, Hazenberg BP, Rapezzi C, Hawkins PN. Nonbiopsy Diagnosis of Cardiac Transthyretin Amyloidosis. Circulation. 2016 Jun 14;133(24):2404-12. doi: 10.1161/CIRCULATIONAHA.116.021612. Epub 2016 Apr 22. PMID 27143678